CLINICAL TRIAL: NCT03558490
Title: Feasibility Assessment of an E-Health System (ZEMY) Designed to Manage Symptoms in Patients With Breast Cancer Under Anti-Cancer Treatment
Brief Title: A Study to Assess the Feasibility of an E-Health System (ZEMY) Designed to Manage Symptoms in Participants With Breast Cancer Under Anti-Cancer Treatment
Acronym: ZEMY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ML39208
Record Dates: First submitted 2018-06-04; First posted 2018-06-15 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ZEMY software (Experimental)
  Interventions: Device: ZEMY software; Drug: Investigator's choice of anti-cancer treatment (except immunotherapy)

INTERVENTIONS:
Device: ZEMY software — The ZEMY software medical device integrates specific algorithms based on international and validated guidelines. It provides individually customized information and defines for the patient an adapted action to follow for each of the following reported symptoms or anti-cancer treatment-related toxicities: diarrhea, fatigue, nausea, vomiting, cutaneous and mucosal toxicities, pain, fever/febrile neutropenia, high blood pressure, anxiety and depression.
  During the 3-month study period, participants will be asked to enter their symptoms among the 10 symptoms listed in ZEMY on their smartphone dedicated to the study. Consequently, ZEMY software will provide to the participants adapted real-time information to advise them on the management of the experienced symptom and recommend hygienic-dietetic advice and symptomatic treatments.
Drug: Investigator's choice of anti-cancer treatment (except immunotherapy) — All anti-cancer treatments (except immunotherapy) will be left to the free choice of investigators. Participants shall be prescribed by the healthcare team both of the following symptomatic treatments: loperamide or any other anti-diarrheic treatment in case of diarrhea; and a prescription for any medication indicated in case of nausea/vomiting. A written prescription will be made by the investigator at screening for loperamide or any other anti-diarrheic treatment and symptomatic treatment for nausea/vomiting with documented dosage and duration.

SUMMARY:
This is a three-month open-label, multicenter, interventional, single arm study located in France, designed to assess feasibility and reliability of the e-Health ZEMY software medical device under investigation for use by participants with breast cancer, who are starting an anti-cancer treatment at any stage of the disease, to manage disease symptoms and anti-cancer treatment-related toxicities while at home.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with breast cancer starting a treatment including oral and/or parenteral anti-cancer drugs (chemotherapy and/or targeted therapies, hormonotherapy)
* Inter-cycle duration between hospital visits ≥14 days (this period of time is estimated to be consistent with a need for support during the home setting period)
* Patients shall be prescribed loperamide or any other anti-diarrheic treatment in case of diarrhea and prescription for any medication indicated in case of nausea/vomiting
* Able to speak and read French and to use a smartphone embedding ZEMY, in the investigator's judgment
* Able to comply with the study protocol, in the investigator's judgment
* Patient affiliated to the national social security or beneficiary to such insurance.

Exclusion Criteria:

* Pregnant
* Already enrolled in a clinical study involving experimental medication or eHealth device
* Concomitant malignancy
* ECOG score >2
* Treated with single hormonotherapy, single surgery or single radiotherapy, immunotherapy.
* Patient whose mental state renders her unable to understand the nature, purposes, and consequences of the study
* Patient not trained to the use of ZEMY
* Patient not trained to take her blood pressure measurement
* Patient deprived of her liberty by judicial or administrative order.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Successfully Use ZEMY | 3 months
  A participant will be considered as successful in terms of the feasibility of using ZEMY if she has completed at least three symptom reported connections and if the rate of completed symptom reported connections for this participant is ≥ 60%.

SECONDARY OUTCOMES:
Percentage of Appropriate Automatic Messages and Recommendations for Each Symptom by ZEMY, as Evaluated by the Investigator at Each Visit | At Weeks 3, 6, 9, and 12 (Up to 3 months)
System Usability Scale Score, Rated by Participants and Healthcare Professionals (HCPs) | At 3 months
Satisfaction with ZEMY, Assessed on a Visual Analog Scale by Participants and HCPs | At 3 months
Percentage of Participant Answered Entries per ZEMY Requests for Solicited Symptom Information | 3 months
Number of Automatic Messages Generated by ZEMY per Participant Over the Study Period | 3 months
Number of Automatic Messages Generated by ZEMY per Symptom Over the Study Period | 3 months
Number of Recommendations Generated by ZEMY per Participant Over the Study Period | 3 months
Number of Recommendations Generated by ZEMY per Symptom Over the Study Period | 3 months
Number and Type of Device Deficiencies | 3 months
  Inadequacy of an investigational medical device related to its identity, quality, durability, reliability, safety or performance. This may include malfunctions, use error, or inadequacy in the information supplied by the manufacturer.
Number and Type of Adverse Device Effects | 3 months
  Adverse event related to the use of an investigational medical device.
Number and Type of Serious Adverse Device Effects | 3 months
  Adverse device effect that has resulted in any of the consequences characteristic of a serious adverse event.
Number and Type of Unanticipated Serious Adverse Device Effects | 3 months
  Serious adverse device effect which by its nature, incidence, severity or outcome has not been identified in the current version of the risk analysis report.
Change From Baseline in the EuroQoL 5-Dimension (EQ-5D-5L) Health Questionnaire Score at Each Study Visit | At Baseline and Weeks 3, 6, 9, and 12 (Up to 3 months)
Change From Baseline in the European Organization for Research and Treatment of Cancer's Quality-of-Life Questionnaire (EORTC QLQ-30) Score at Each Study Visit | At Baseline and Weeks 3, 6, 9, and 12 (Up to 3 months)
Change From Baseline in the European Organization for Research and Treatment of Cancer's Breast Cancer-Specific Quality-of-Life Questionnaire (EORTC QLQ-BR23) Score at Each Study Visit | At Baseline and Weeks 3, 6, 9, and 12 (Up to 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- France (5):
  - Centre Francois Baclesse; Oncologie, Caen
  - Centre Jean Perrin; Oncologie, Clermont-Ferrand
  - Hopital Prive Jean Mermoz; Cancerologie, Lyon
  - Hopital Saint Louis; Oncologie Medicale, Paris
  - Institut du Cancer Coulancy Reims, Reims